CLINICAL TRIAL: NCT01819987
Title: Home-based & Technology-centered Childhood Obesity Prevention for Mothers With Young Children
Brief Title: HomeTech Healthy Lifestyle Program for Mothers With Young Children
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HomeTech healthy lifestyle
Record Dates: First submitted 2013-03-18; First posted 2013-03-28 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Overweight
Keywords: Overweight; mother; childhood obesity prevention; Chinese American
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Intervention Model Description: A randomized, controlled study was used. The intervention group received tablet based intervention and the control group received printed health information relevant to preschool-aged children in Chinese over the eight weeks.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants, investigator and outcome assessor were blinded to the group assignment.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mailing information (Active Comparator): Participants in the mailing information group will receive general health promotion topics relevant to preschool-age children (such as immunization, injury prevention and school readiness) via mailing materials that are bilingual weekly for eight weeks. These materials will be obtained from CDC and AAP.
  Interventions: Behavioral: Mailing information
- Tablet computer (Experimental): Participants in the intervention group will receive eight weekly online sessions and interactive activities delivered through tablet computers. Intervention participants will receive instructions for accessing the program via the tablet at an in-person session. Automated weekly emails will be sent to participating mothers for the intervention duration to encourage study engagement.
  Interventions: Behavioral: Tablet computer

INTERVENTIONS:
Behavioral: Tablet computer — Participants in the intervention group will receive eight weekly online sessions and interactive activities delivered through tablet computers. Intervention participants will receive instructions for accessing the program via the tablet at an in-person session. Automated weekly emails will be sent to participating mothers for the intervention duration to encourage study engagement.
  Arms: Tablet computer
Behavioral: Mailing information — Participants in the control group will receive general health promotion topics relevant to preschool-age children (such as immunization, injury prevention and school readiness) via mailing materials that are bilingual weekly for eight weeks. These materials will be obtained from CDC and AAP.
  Arms: Mailing information

SUMMARY:
About 17% of Chinese American preschool children are obese, compared to 12.4%of all children from age three to five years residing in the US; the prevalence of obesity is expected to increase in the future. Therefore, the proposed study will adapt a home-based and technology-centered childhood obesity prevention program for low-income Chinese American mothers of children three to five years old. The aims of the study are to assess the feasibility of the intervention and estimate the effect sizes on children's and mothers' outcomes.

DETAILED DESCRIPTION:
This study aims to adapt and implement a family-centered and technology-based intervention to prevent obesity in young Chinese American children from low-income families with overweight mothers. The proposed study framework is based on the Information Motivation Behavioral Skills Model, which includes the mothers' gained knowledge/information, increased personal and social motivators, and acquired behavioral skills towards behavioral changes. The intervention will be developed with a Community Advisory Committee and validated for cultural appropriateness through a beta-testing process. The validated intervention will be implemented thereafter. Eligible overweight mothers with young Chinese American children (ages three to five years) will be recruited from local day care settings, low-income housing and Head Start programs to participate in the study. Participants will be randomized into either the intervention (N=15) or control group (N=15). Participants in the intervention group will receive the 8-week online interactive sessions and activities delivered through tablet computers. Participants in the control group will receive general health promotion topics relevant to preschool-age children via mailing materials weekly for eight weeks.

ELIGIBILITY:
Inclusion Criteria:

* Children:
* must be between ages three and five
* have a mother who identifies her child as Chinese;
* be healthy-defined as free of chronic or acute illness.
* Mothers:
* must identify themselves as Chinese
* the primary provider of the child,
* be able to speak and read Chinese or English;
* with a BMI >= 23.0;
* meet low-income requirements in the Bay Area.

Exclusion Criteria:

* Have acute or chronic conditions that prevent performing daily activities

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2016-06-01 (Actual); Study Completion 2016-06-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline body mass index at 5 months | Baseline and at 5 months
  Participants will have their weight and height measured and body mass index will be calculated. Change of BMI from baseline will be assessed at 5 months post baseline

SECONDARY OUTCOMES:
Change from baseline physical activity at 2 months | Baseline and 2 months
  Participants will wear Actigraphy for 7 days at baseline and at 2 months. Change of physical activity from baseline will be assessed at 2 months post baseline.
Change from Baseline Sedentary activity at 2 months | baseline and 2 months
  Participants will complete Family Eating and Activity Habits Questionnaire at baseline and at 2 month.
Change from Baseline Parental Feeding Practice at 2 months | baseline and 2 months
  Participants will complete Child Feeding Questionnaire at baseline and at 2 months . Change of parental feeding practice from baseline will be assessed at 2 months.
Change from Baseline Self-efficacy regarding diet and physical activity at 2 months | baseline and 2 months
  Participants will complete self-efficacy questionnaire regarding nutrition and physical behavior at baseline and at 2 months. Change of self-efficacy from baseline will be assessed at 2 months.
Change from baseline physical activity level at 5 months | Baseline and 5 months
  Change in baseline physical actiivty level will be measured at 5 months.
Change from Baseline Sedentary activity at 5 months | baseline and 5 months
  Participants will complete Family Eating and Activity Habits Questionnaire at baseline and at 5 months.
Change from Baseline Parental Feeding Practice at 5 months | baseline and 5 months
  Participants will complete Child Feeding Questionnaire at baseline and at 5 months . Change of parental feeding practice from baseline will be assessed at 5 months.
Change from Baseline Self-efficacy regarding diet and physical activity at 5 months | baseline and 5 months
  Participants will complete self-efficacy questionnaire regarding nutrition and physical behavior at baseline and at 5 months. Change of self-efficacy from baseline will be assessed at 5 months.

CONTACTS AND LOCATIONS:
Overall Officials: Jyu-Lin Chen, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States